CLINICAL TRIAL: NCT01523691
Title: Repeating Patterns of Sleep Restriction and Recovery - do we Get Used to it?
Brief Title: Repeating Patterns of Sleep Restriction and Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Monika Haack, Assistant Professor of Neurology, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2010P000399; R01HL105544-01A1 (NIH)
Record Dates: First submitted 2011-11-30; First posted 2012-02-01 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Healthy
Keywords: Healthy individuals
MeSH Terms: interventions — Salvage Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- repeated sleep restriction and recovery (Experimental)
  Interventions: Behavioral: Repeated sleep restriction and recovery
- control sleep (Experimental)
  Interventions: Behavioral: Control sleep

INTERVENTIONS:
Behavioral: Repeated sleep restriction and recovery — Repeated cycles of sleep restriction and sleep recovery
  Arms: repeated sleep restriction and recovery
Behavioral: Control sleep — Regular amounts of sleep across study protocol
  Arms: control sleep

SUMMARY:
Goal of this study is to test the hypothesis that repeated exposure to cycles of insufficient sleep increases susceptibility to a variety of disease states by progressively compromising the integrity of stress response systems.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18.5 and 30 kg/m2
* For female participants: regular menstrual cycles
* Daily sleep duration in the normal range
* Blood chemistry in the normal range

Exclusion Criteria:

* Active infection/disease
* History of psychiatric, neurological, pain-related, immune, or cardiovascular disease; significant allergy
* Pregnant/nursing
* Respiratory disturbance index of >5 events/hour on polysomnographic sleep study, leg movements with arousal >10/hour; sleep efficiency <80%
* Regular medication use other than oral contraceptives
* Donation of blood or platelets 3 month prior to or in-between study arms

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2011-08; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
stress-related markers | Participants will be followed for the duration of hospital stay, an axpected average of 2 x 25 days.
  cortisol, ACTH, norepinephrine, IL-6, COX in blood/urine, among others

SECONDARY OUTCOMES:
subjective stress-related markers | Participants will be followed for the duration of hospital stay, an axpected average of 2 x 25 days.
  Computerized rating scales for the assessment of physical and emotional well-being

CONTACTS AND LOCATIONS:
Overall Officials: Monika Haack, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States